CLINICAL TRIAL: NCT04610502
Title: Randomized, Controlled, Double-blind, Multicenter Clinical Study to Compare the Efficacy and Safety of the Administration of Two Hyperimmune Equine Anti-Sars-CoV-2 ("S" and "M") Serum Formulations in Hospitalized Patients With COVID-19
Brief Title: Efficacy and Safety of Two Hyperimmune Equine Anti Sars-CoV-2 Serum in COVID-19 Patients
Acronym: SECR-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Caja Costarricense de Seguro Social (Other Government)
Collaborators: Universidad de Costa Rica (Other); Ministry of Health Costa Rica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R020-SABI-00259
Record Dates: First submitted 2020-09-15; First posted 2020-10-30 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: COVID-19; Anti-SARS-CoV-2 Equine Immunoglobulin; Passive Immunotherapy; Neutralizing Equine Antibodies.
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equine immunoglobulin anti SARS-CoV-2 formulation S (Experimental): Experimental equine Imunoglobulins antiSARSCov" Formuation S
  Interventions: Biological: Administration of Equine immunoglobulin anti SARS-CoV-2
- Equine immunoglobulin anti SARS-CoV-2 formulation M (Experimental): Experimental equine Imunoglobulins antiSARSCov" Formuation M
  Interventions: Biological: Administration of Equine immunoglobulin anti SARS-CoV-2

INTERVENTIONS:
Biological: Administration of Equine immunoglobulin anti SARS-CoV-2 — The participants will receive premedication with Acetaminophen 500mg PO, Cimetidine300mg IV and Chlortrimeton 10mg IV. Then the investigators will do the Administration of Equine Imunoglobulin anti SARS Cov 2 on day 1 a vial of 10ml of the drug during 1 hour Intravenously. Then the hospitalized participants will be followed until they are discharged.

SUMMARY:
Reports of the use of plasma from convalescent patients and purified immunoglobulin preparations in respiratory infections by various viral agents and SARS-CoV-2 in severely ill patients suggest that specific neutralizing antibodies may benefit their clinical course. During the previous SARS-CoV epidemic in 2003, preparations of hyperimmune equine serum were produced and demonstrated in vitro viral neutralization. These preparations were also successful in several animal models. Taking advantage of the important trajectory of our country in the study and use of equine hyperimmune serums with neutralizing antibodies for snake venom, preparations of hyperimmune serums against recombinant proteins of SARS-CoV-2 were produced through repeated immunization of horses, a first group of animals was inoculated with the "S" (Spike) protein of the virus and the second group with a mixture "M" of the S1 (Spike) proteins, the N (Nucleoprotein) protein and a construct with epitopes of the S1, E (Envelope) and M (Membrane) proteins, generating two different pharmaceutical preparations.

Objective: Evaluate the efficacy and safety of two hyperimmune equine serum anti-Sars-CoV-2 ("S" and "M") formulations as an addition to the standard therapeutic approach for hospitalized patients with COVID-19 over 18 years of age with the presence of at least 2 risk factors and a symptom onset period not exceeding 10 days.

A total of 52 patients will be included and randomly divided into two balanced groups. On day 1, all participants from each group will receive an intravenous infusion containing 10ml (one vial) of hyperimmune equine anti-Sars-CoV-2 serum labeled as A or B.

Patients will be evaluated clinically, general laboratory, SARS-CoV-2 serologies, SARS-CoV-2 viral load and cytokines level as well as pulmonary ultrasound. Data will be collected for both groups on Days 0 to 7, 10 and 14 or discharge after completion of treatment. The study will end for each participant on the day of discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the study by signing the prior informed consent.
* Age over 18 years.
* Inpatient with RT-PCR confirmation of SARS-CoV-2.
* Period of onset of symptoms related to COVID-19 not greater than 10 days
* Presence of at least 2 documented risk factors
* Moderate and severe clinical presentation of the disease.

Exclusion Criteria:

* Patients who did not sign the Informed Consent.
* Critical patient.
* Patient previously bitten by a snake that was treated with equine hyperimmune serum.
* Patients with COVID-19 on an outpatient basis.
* Pregnant women.
* Patients in Hemodialysis program.
* Patients who have already received plasma from a convalescent COVID-19 patient.
* Patients who were classified prior to the diagnosis of COVID-19 by the treating physician as having a reserved prognosis with a short lifespan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-06 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of two formulations of equine anti-SARS-CoV-2 immunoglobulins ("S" and "M"). | 2,3,4,5,7,10,14 Days
  Change in clinical status (days requiring supplemental oxygen) between the two treatment groups.
To evaluate safety of two formulations of equine anti-SARS-CoV-2 immunoglobulins ("S" and "M"). | 3 months
  To identify the adverse effects of anti-Sars-CoV-2 type "S" or type "M" equine immunoglobulins administered to patients diagnosed as SARS-CoV-2 positive, with the presence of at least 2 risk factors and a symptom onset period of no more than 10 days.

SECONDARY OUTCOMES:
Viral load | Days 2,3,4,5,7,10,14
  Change of viral load (number of copies of SARS Cov2 per ml)
Mortality | days 14, 24
  Change in mortality between the two treatment groups.
Hospital stay | Day 14, 24
  Change in the overall hospital stay of patients between the two treatment groups.
ventilatory support | Day 24
  Change in duration of ventilation support in the two treatment groups
blood levels of immunoglobulins against SARS-CoV-2 | Days 2,3,4,5,7,10,14
  Change in titer of immunoglobulins blood levels (UA/ml) against SARS-CoV-2 between the two treatment groups.
inflammatory markers | day 10
  Rate of virologic clearance by nasopharyngeal swab at day 10
thrombotic marker levels | days 2, 3, 4, 7, 10, and 14
  7. Difference in the decrease of thrombotic marker levels (D-dimer, fibrinogen, prothrombin time, TTP) on study days 2, 3, 4, 7, 10, and 14 or at discharge between the two treatment groups
negativization period of RT-PCR on nasopharyngeal swabbing (Reverse transcription polymerase chain reaction) | 1 month
  8. Difference in the number of days elapsed between two negative determinations separated by at least 24 hours in the COVID-19 test by RT-PCR on nasopharyngeal swabbing between the two treatment groups
SpFI (Partial saturation Oxigen/inspired fraction of Oxigen) gain | Days 2,3,4,5,7,10,14
  Improvement in SAFI (SatO2/FiO2) between the two treatment groups.
Lung Ultrasound | days 3,10
  Change in POCUS score between the two treatment groups. (Minimum: 0 = normal; Maximum: 32= Multiple Lungs Consolidations).
Adverse events | days 2,3,4,5,6,7,10,14,24
  Number of adverse events as measured by CTCAE v. 5.0 between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Sanabria, PhD, Principal Investigator — Caja Costarricense de Seguro Social; Willem Bujan, MBA, Study Chair — UCR
Locations (4):
- Costa Rica (4):
  - Centro Especializado de Atención COVID19 (CEACO), San José
  - Hospital Dr. Rafael Ángel Calderón Guardia, San José
  - Hospital México, San José
  - Hospital San Juan de Dios, San José

IPD SHARING:
Plan to Share IPD: No